CLINICAL TRIAL: NCT03332771
Title: A 52-week Randomized, Double-blind, Double-dummy, Active and Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Efficacy and Safety of Sotagliflozin Compared to Glimepiride or Placebo Added to Metformin in Patients With Type 2 Diabetes Who Have Inadequate Glycemic Control With Metformin Monotherapy
Brief Title: Efficacy and Safety of Sotagliflozin Versus Glimepiride and Placebo in Participants With Type 2 Diabetes Mellitus That Are Taking Metformin Monotherapy
Acronym: SOTA-GLIM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC14838; 2016-001801-17 (EudraCT Number); U1111-1190-7596 (Other: UTN)
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol; glimepiride; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sotagliflozin 400 mg (Experimental): Following a 2-week run-in period, two Sotagliflozin 200 mg, tablets, and two Glimepiride-matching placebo capsules, taken orally once daily before the first meal of the day in the double-blind treatment period up to 52 weeks.
  Interventions: Drug: Sotagliflozin (SAR439954); Drug: Metformin; Drug: Placebo
- Sotagliflozin 200 mg (Experimental): Following a 2-week run-in period, one Sotagliflozin 200 mg, tablet and one Sotagliflozin-matching placebo tablet, and two Glimepiride-matching placebo capsules, taken orally once daily before the first meal of the day in the double-blind treatment period up to 52 weeks.
  Interventions: Drug: Sotagliflozin (SAR439954); Drug: Metformin; Drug: Placebo
- Glimepiride (Active Comparator): Following a 2-week run-in period, two Sotagliflozin-matching placebo tablets, and combination of two Glimepiride capsules with adequate dose strengths per dose titration (titrated up to 6mg), taken orally once daily before the first meal of the day in the double-blind treatment period up to 52 weeks.
  Interventions: Drug: Glimepiride; Drug: Metformin; Drug: Placebo
- Placebo (Placebo Comparator): Following a 2-week run-in period, two Sotagliflozin-matching placebo tablets and two Glimepiride-matching placebo capsules, taken orally once daily before the first meal of the day in the double-blind treatment period up to 52 weeks.
  Interventions: Drug: Metformin; Drug: Placebo

INTERVENTIONS:
Drug: Sotagliflozin (SAR439954) — Pharmaceutical form: tablet
  Route of administration: oral
  Arms: Sotagliflozin 200 mg; Sotagliflozin 400 mg
Drug: Glimepiride — Pharmaceutical form: capsule
  Route of administration: oral
  Arms: Glimepiride
Drug: Metformin — Pharmaceutical form: tablet
  Route of administration: oral
Drug: Placebo — Pharmaceutical form: tablet
  Route of administration: oral
  Arms: Glimepiride; Placebo; Sotagliflozin 200 mg
Drug: Placebo — Pharmaceutical form: capsule
  Route of administration: oral
  Arms: Placebo; Sotagliflozin 200 mg; Sotagliflozin 400 mg

SUMMARY:
Primary Objective:

To demonstrate the non-inferiority of Sotagliflozin 400 milligrams (mg) compared to Glimepiride on hemoglobin A1c (HbA1c) reduction at Week 52 in participants with Type 2 Diabetes (T2D) who have inadequate glycemic control with metformin.

Secondary Objectives:

To demonstrate the superiority of Sotagliflozin 400 mg compared to Glimepiride on change in body weight, systolic blood pressure (SBP) in participants with baseline SBP ≥130 millimeter of mercury (mmHg), SBP in all participants, and proportion of participants with at least 1 documented symptomatic hypoglycemic event (≤70 milligrams per deciliter [mg/dL]).

* To demonstrate the superiority of Sotagliflozin 400 mg compared to placebo on change in HbA1c, body weight, SBP in participants with baseline SBP ≥130 mmHg, SBP in all participants.
* To demonstrate the superiority of Sotagliflozin 200 mg compared to placebo on change in HbA1c.
* To demonstrate the non-inferiority of Sotagliflozin 400 mg compared to Glimepiride on change in HbA1c.
* To demonstrate the superiority of Sotagliflozin 400 mg compared to Glimepiride on change in HbA1c.
* To evaluate the safety and tolerability of Sotagliflozin compared to Glimepiride and placebo.

DETAILED DESCRIPTION:
Up to 58 weeks, including a Screening Period consisting of a Screening phase of up to 2 weeks, a 2-week single-blind placebo Run-in phase, a 52-week double-blind Treatment Period, and a 2-week post-treatment Follow-up period to collect safety information.

ELIGIBILITY:
Inclusion criteria :

* Participants with Type 2 Diabetes (T2D) treated with metformin at a stable dose ≥1500 milligrams per day (mg/day) or maximum tolerated dose (documented) for at least 12 weeks prior to Screening Visit; in case of documented lack of tolerance, metformin dose <1500 mg/day is acceptable, and the dose should be stable for at least 12 weeks prior to Screening Visit.
* Participants has given written informed consent to participate in the study in accordance with local regulations.

Exclusion criteria:

* Age <18 years at the Screening Visit or <legal age of majority, whichever is greater.
* Type 1 diabetes mellitus.
* HbA1c, HbA1c <7.0% or HbA1c >10% at Screening.
* Fasting Plasma Glucose (FPG) >15 millimoles per liter (mmol/L) (>270 milligram per deciliter [mg/dL]) measured by the central laboratory at Screening (Visit 1) and confirmed by a repeat test (>15 mmol/L [>270 mg/dL]) before randomization.
* Body mass index ≤20 or >45 kilogram per meter square (kg/m^2) at Screening.
* Pregnant (confirmed by pregnancy test at the Screening) or breast-feeding women.
* Women of childbearing potential (WOCBP) not willing to use highly effective method(s) of birth control during the study treatment period and the follow-up period, or who are unwilling or unable to be tested for pregnancy (see Appendix A) during the study.
* Previous use of any antidiabetic drug other than Metformin within 12 weeks preceding the Screening Visit.
* Use of a selective Sodium-glucose co-transporter-2 (SGLT2) inhibitor (e.g., Canagliflozin, Dapagliflozin, or Empagliflozin) within 3 months prior to the Screening visit.
* Use of systemic glucocorticoids (excluding topical, or ophthalmic application, intra-articular, nasal spray or inhaled forms) for more than 10 consecutive days within 90 days prior to the Screening Visit.
* Previous insulin use >1 month (at any time, except for treatment of gestational diabetes).
* History of prior gastric surgical procedure, including gastric banding, or inflammatory bowel disease within 3 years prior to the Screening Visit.
* Difficulty swallowing such that the participants cannot take the investigational medicinal product (IMP).
* History of diabetic ketoacidosis or nonketotic hyperosmolar coma within 12 weeks prior to the Screening Visit.
* Mean of 3 separate blood pressure measurements >180 millimeter of mercury (mmHg) (SBP) or >100 mmHg (DBP).
* History of hypertensive emergency within 12 weeks prior to Screening.
* Participants who have previously been randomized in any clinical trial of Sotagliflozin/LX4211.
* Participants with severe renal disease as defined by an estimated glomerular filtration rate (eGFR) of <30 milliliter per minute per meter square (mL/min/1.73 m^2) at Screening, based on the 4 variable Modification of Diet in Renal Disease (MDRD) equation (or according to the renal function restrictions of metformin use defined in the local approved label).
* Participants with severe anemia, severe cardiovascular (including congestive heart failure New York Heart Association IV), respiratory, hepatic, neurological, psychiatric, or active malignant tumor or other major systemic disease that, according to Investigator, will preclude their safe participation in this study, or will make implementation of the protocol or interpretation of the study results difficult.
* Aspartate aminotransferase and/or alanine aminotransferase: >3 times the upper limit of the normal laboratory range (ULN).
* Total bilirubin: >1.5 times ULN (except in case of Gilbert's syndrome).
* Participants who have taken other investigational drugs within 12 weeks or 5 half-lives from Screening whichever is longer.
* Participants unwilling or unable to perform self-monitoring blood glucose (SMBG), complete the participant diary, or comply with study visits and other study procedures as required per protocol.
* Participants with contraindication to glimepiride as per local labelling.
* Participants with contraindication to metformin as per local labelling.

The above information is not intended to contain all considerations relevant to a Participants potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 954 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suman Wason, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (142):
- United States (115):
  - Investigational Site Number 8407040, Birmingham, Alabama
  - Investigational Site Number 8407048, Birmingham, Alabama
  - Investigational Site Number 8407035, Little Rock, Arkansas
  - Investigational Site Number 8407051, Anaheim, California
  - Investigational Site Number 8407065, Canoga Park, California
  - Investigational Site Number 8407078, Carmichael, California
  - Investigational Site Number 8407089, Downey, California
  - Investigational Site Number 8407011, Gold River, California
  - Investigational Site Number 8407044, Greenbrae, California
  - Investigational Site Number 8407006, Huntington Park, California
  - Investigational Site Number 8407037, Lemon Grove, California
  - Investigational Site Number 8407100, Lomita, California
  - Investigational Site Number 8407033, Long Beach, California
  - Investigational Site Number 8407019, Los Angeles, California
  - Investigational Site Number 8407098, Northridge, California
  - Investigational Site Number 8407094, Norwalk, California
  - Investigational Site Number 8407106, Pomona, California
  - Investigational Site Number 8407096, Rancho Cucamonga, California
  - Investigational Site Number 8407036, Sacramento, California
  - Investigational Site Number 8407084, Tarzana, California
  - Investigational Site Number 8407034, Upland, California
  - Investigational Site Number 8407032, Van Nuys, California
  - Investigational Site Number 8407004, Walnut Creek, California
  - Investigational Site Number 8407117, Wildomar, California
  - Investigational Site Number 8407045, Colorado Springs, Colorado
  - Investigational Site Number 8407074, Bradenton, Florida
  - Investigational Site Number 8407027, Clearwater, Florida
  - Investigational Site Number 8407103, Cooper City, Florida
  - Investigational Site Number 8407021, Coral Gables, Florida
  - Investigational Site Number 8407062, Lake Worth, Florida
  - Investigational Site Number 8407121, Ocoee, Florida
  - Investigational Site Number 8407024, Orlando, Florida
  - Investigational Site Number 8407038, Palmetto Bay, Florida
  - Investigational Site Number 8407093, Pembroke Pines, Florida
  - Investigational Site Number 8407107, Spring Hill, Florida
  - Investigational Site Number 8407091, Tampa, Florida
  - Investigational Site Number 8407113, Tampa, Florida
  - Investigational Site Number 8407092, West Palm Beach, Florida
  - Investigational Site Number 8407115, Winter Haven, Florida
  - Investigational Site Number 8407017, Chicago, Illinois
  - Investigational Site Number 8407018, Elgin, Illinois
  - Investigational Site Number 8407046, Gurnee, Illinois
  - Investigational Site Number 8407119, Springfield, Illinois
  - Investigational Site Number 8407075, Waterloo, Iowa
  - Investigational Site Number 8407120, West Des Moines, Iowa
  - Investigational Site Number 8407095, Topeka, Kansas
  - Investigational Site Number 8407083, Wichita, Kansas
  - Investigational Site Number 8407043, Lexington, Kentucky
  - Investigational Site Number 8407087, Lexington, Kentucky
  - Investigational Site Number 8407060, Lake Charles, Louisiana
  - Investigational Site Number 8407058, New Orleans, Louisiana
  - Investigational Site Number 8407009, New Orleans, Louisiana
  - Investigational Site Number 8407079, Zachary, Louisiana
  - Investigational Site Number 8407085, Baltimore, Maryland
  - Investigational Site Number 8407001, Rockville, Maryland
  - Investigational Site Number 8407069, Troy, Michigan
  - Investigational Site Number 8407110, Olive Branch, Mississippi
  - Investigational Site Number 8407054, Bridgeton, Missouri
  - Investigational Site Number 8407049, Norfolk, Nebraska
  - Investigational Site Number 8407039, Omaha, Nebraska
  - Investigational Site Number 8407061, Papillion, Nebraska
  - Investigational Site Number 8407108, Las Vegas, Nevada
  - Investigational Site Number 8407050, Albuquerque, New Mexico
  - Investigational Site Number 8407116, New York, New York
  - Investigational Site Number 8407086, New York, New York
  - Investigational Site Number 8407122, New York, New York
  - Investigational Site Number 8407123, West Seneca, New York
  - Investigational Site Number 8407020, Greensboro, North Carolina
  - Investigational Site Number 8407114, Lenoir, North Carolina
  - Investigational Site Number 8407015, Morehead City, North Carolina
  - Investigational Site Number 8407030, Salisbury, North Carolina
  - Investigational Site Number 8407041, Wilmington, North Carolina
  - Investigational Site Number 8407101, Winston-Salem, North Carolina
  - Investigational Site Number 8407099, Cincinnati, Ohio
  - Investigational Site Number 8407081, Lyndhurst, Ohio
  - Investigational Site Number 8407057, Norman, Oklahoma
  - Investigational Site Number 8407073, Oklahoma City, Oklahoma
  - Investigational Site Number 8407068, Eugene, Oregon
  - Investigational Site Number 8407104, Beaver, Pennsylvania
  - Investigational Site Number 8407025, Hatboro, Pennsylvania
  - Investigational Site Number 8407053, Lansdale, Pennsylvania
  - Investigational Site Number 8407016, Charleston, South Carolina
  - Investigational Site Number 8407071, Greer, South Carolina
  - Investigational Site Number 8407022, Mt. Pleasant, South Carolina
  - Investigational Site Number 8407031, Mt. Pleasant, South Carolina
  - Investigational Site Number 8407014, Jefferson City, Tennessee
  - Investigational Site Number 8407002, Knoxville, Tennessee
  - Investigational Site Number 8407056, Memphis, Tennessee
  - Investigational Site Number 8407026, Austin, Texas
  - Investigational Site Number 8407029, Beaumont, Texas
  - Investigational Site Number 8407070, Carrollton, Texas
  - Investigational Site Number 8407102, Corpus Christi, Texas
  - Investigational Site Number 8407023, Dallas, Texas
  - Investigational Site Number 8407111, Dallas, Texas
  - Investigational Site Number 8407013, Fort Worth, Texas
  - Investigational Site Number 8407080, Houston, Texas
  - Investigational Site Number 8407088, Houston, Texas
  - Investigational Site Number 8407090, Katy, Texas
  - Investigational Site Number 8407042, Lampasas, Texas
  - Investigational Site Number 8407067, Lufkin, Texas
  - Investigational Site Number 8407118, Lufkin, Texas
  - Investigational Site Number 8407059, McAllen, Texas
  - Investigational Site Number 8407012, Mesquite, Texas
  - Investigational Site Number 8407007, Plano, Texas
  - Investigational Site Number 8407005, San Antonio, Texas
  - Investigational Site Number 8407064, San Antonio, Texas
  - Investigational Site Number 8407010, Schertz, Texas
  - Investigational Site Number 8407076, Splendora, Texas
  - Investigational Site Number 8407063, Clinton, Utah
  - Investigational Site Number 8407055, Holladay, Utah
  - Investigational Site Number 8407097, Ogden, Utah
  - Investigational Site Number 8407072, Salt Lake City, Utah
  - Investigational Site Number 8407124, Manassas, Virginia
  - Investigational Site Number 8407105, Richmond, Virginia
  - Investigational Site Number 8407028, Renton, Washington
- Bulgaria (9):
  - Investigational Site Number 1007002, Gabrovo
  - Investigational Site Number 1007008, Plovdiv
  - Investigational Site Number 1007003, Plovdiv
  - Investigational Site Number 1007001, Rousse
  - Investigational Site Number 1007004, Smolyan
  - Investigational Site Number 1007009, Sofia
  - Investigational Site Number 1007005, Stara Zagora
  - Investigational Site Number 1007006, Stara Zagora
  - Investigational Site Number 1007007, Varna
- Hungary (8):
  - Investigational Site Number 3487005, Balatonfüred
  - Investigational Site Number 3487001, Budapest
  - Investigational Site Number 3487010, Budapest
  - Investigational Site Number 3487006, Debrecen
  - Investigational Site Number 3487008, Debrecen
  - Investigational Site Number 3487002, Kecskemét
  - Investigational Site Number 3487004, Nyíregyháza
  - Investigational Site Number 3487007, Nyíregyháza
- Slovakia (10):
  - Investigational Site Number 7037004, Bardejov
  - Investigational Site Number 7037008, Bratislava
  - Investigational Site Number 7037007, Bratislava
  - Investigational Site Number 7037005, Košice
  - Investigational Site Number 7037002, Levice
  - Investigational Site Number 7037010, Nitra
  - Investigational Site Number 7037009, Rožňava
  - Investigational Site Number 7037001, Sabinov
  - Investigational Site Number 7037003, Trnava
  - Investigational Site Number 7037006, Vrútky

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) and supporting clinical documents are available for request at clinicalstudydatarequest.com. While making information available Sanofi continues to protect the privacy of the participants in clinical trials and to remove commercially confidential information (CCI). Details on Data Sharing criteria and process for requesting access can be found at this web address: clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 138 investigative sites in United States, Bulgaria, Hungary, and Slovakia from 01 December 2017 to 06 September 2019.
Pre-assignment Details: Participants with diagnosis of Type 2 Diabetes Mellitus were enrolled in 1 of 4 treatment groups: Placebo or Sotagliflozin 200 mg or Sotagliflozin 400 mg or Glimepiride. Participants were randomly assigned in the ratio of 1:1:2:2 to these reporting groups. Total of 954 participants were enrolled in study, out of which 952 were randomized and treated.
Period: Overall Study
Arm/Group | Placebo | Sotagliflozin 400 mg | Sotagliflozin 200 mg | Glimepiride
Started | 159 | 317 | 160 | 318
Completed | 125 | 266 | 128 | 270
Not Completed | 34 | 51 | 32 | 48
Not completed — Adverse Event | 6 | 4 | 1 | 3
Not completed — Poor Compliance to Protocol | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 2 | 2 | 1 | 2
Not completed — At the Participant's own request | 20 | 26 | 14 | 23
Not completed — Reason Not Specified | 6 | 18 | 16 | 19

BASELINE CHARACTERISTICS:
Population: The randomized population included any participant who had been allocated to a randomized treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sotagliflozin 400 mg | Sotagliflozin 200 mg | Glimepiride | Total
Number analyzed (Participants) | 159 | 317 | 160 | 318 | 954
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (11.2) | 59.7 (10.4) | 58.6 (9.9) | 59.8 (9.6) | 59.4 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 157 | 75 | 143 | 452
  Male | 82 | 160 | 85 | 175 | 502
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 48 | 85 | 53 | 111 | 297
  Not Hispanic or Latino | 110 | 230 | 106 | 207 | 653
  Unknown or Not Reported | 1 | 2 | 1 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1 | 2
  Asian | 3 | 5 | 3 | 4 | 15
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2 | 0 | 4
  Black or African American | 13 | 34 | 19 | 36 | 102
  White | 141 | 269 | 136 | 277 | 823
  More than one race | 1 | 3 | 0 | 0 | 4
  Unknown or Not Reported | 0 | 4 | 0 | 0 | 4
Region of Enrollment [Number; unit: participants]
  Bulgaria | 7 | 17 | 5 | 16 | 45
  Hungary | 22 | 48 | 24 | 42 | 136
  Slovakia | 12 | 28 | 10 | 30 | 80
  United States | 118 | 224 | 121 | 230 | 693
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percentage of HbA1c] | 8.12 (0.73) | 8.09 (0.78) | 8.11 (0.86) | 8.07 (0.79) | 8.09 (0.79)
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: millimeter of mercury (mmHg)] | 133.23 (14.90) | 133.17 (14.37) | 132.78 (13.29) | 134.66 (14.43) | 133.61 (14.30)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c at Week 52
Description: An analysis of covariance (ANCOVA) model was used for the analysis.
Time Frame: Baseline, Week 52
Population: Intend to treat (ITT) population included all randomized participants. Missing data are imputed using the retrieved dropouts imputation method.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | Sotagliflozin 400 mg | Sotagliflozin 200 mg | Glimepiride
Number analyzed (Participants) | 159 | 317 | 160 | 318
percentage of HbA1c | -0.40 (0.187) | -0.65 (0.101) | -0.49 (0.114) | -0.61 (0.093)
Statistical Analysis 1: Comparison: Sotagliflozin 400 mg vs Glimepiride; The change from baseline to Week 52 is analyzed using ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of SBP (<130, ≥130 mmHg) at screening, and country as fixed effects, and baseline HbA1c as a covariate; Test type: Non-Inferiority — The non-inferiority hypothesis was declared significant if the upper bound of the 2-sided 95% confidence interval (CI) for the adjusted mean difference is <0.3; p = 0.3306, ANCOVA; Difference in Least Squares (LS) Mean = 0.12, 95% CI 2-sided [-0.120 to 0.357], Standard Error of Mean 0.122
Statistical Analysis 2: Comparison: Sotagliflozin 200 mg vs Glimepiride; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — The non-inferiority hypothesis was declared significant if the upper bound of the 2-sided 95% CI for the adjusted mean difference is <0.3; p = 0.7112, ANCOVA; Difference in LS Mean = -0.04, 95% CI 2-sided [-0.265 to 0.181], Standard Error of Mean 0.114

2. Secondary Outcome: Change From Baseline in Hemoglobin A1c at Week 26
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline, Week 26
Population: ITT population included all randomized participants. Missing data are imputed using the washout imputation method.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | Sotagliflozin 400 mg | Sotagliflozin 200 mg | Glimepiride
Number analyzed (Participants) | 159 | 317 | 160 | 318
percentage of HbA1c | -0.41 (0.097) | -0.77 (0.076) | -0.61 (0.098) | -1.02 (0.075)
Statistical Analysis 1: Comparison: Sotagliflozin 400 mg vs Glimepiride; The change from baseline to Week 26 is analyzed using ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of SBP (<130, ≥130 mmHg) at screening, and country as fixed effects, and baseline HbA1c as a covariate; Test type: Superiority; p = 0.0827, ANCOVA; Difference in LS Mean = -0.21, 95% CI 2-sided [-0.440 to 0.027], Standard Error of Mean 0.119
Statistical Analysis 2: Comparison: Sotagliflozin 200 mg vs Glimepiride; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0003, ANCOVA; Difference in LS Mean = -0.37, 95% CI 2-sided [-0.571 to -0.167], Standard Error of Mean 0.103

3. Secondary Outcome: Change From Baseline in Body Weight at Week 26 and 52
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline, Week 26, Week 52
Population: ITT population included all randomized participants. Missing data are imputed using the retrieved dropouts & washout imputation method.
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | Placebo | Sotagliflozin 400 mg | Sotagliflozin 200 mg | Glimepiride
Number analyzed (Participants) | 159 | 317 | 160 | 318
kilogram (kg)
  Change at Week 26 | -1.26 (0.329) | -2.75 (0.257) | -2.24 (0.336) | 0.70 (0.256)
  Change at Week 52 | -0.47 (1.406) | -2.64 (0.503) | -1.74 (0.707) | 0.94 (0.452)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 400 mg; The change from baseline to Week 26 is analyzed using ANCOVA model with treatment groups (placebo, sotagliflozin 200 mg, sotagliflozin 400 mg, glimepiride), randomization strata of HbA1c (≤ 8.5, >8.5%) at screening, randomization strata of SBP (<130,≥ 130 mmHg) at screening, and country as fixed effects, and baseline body weight as a covariate; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LS Mean = -1.49, 95% CI 2-sided [-2.173 to -0.803], Standard Error of Mean 0.349
Statistical Analysis 2: Comparison: Sotagliflozin 400 mg vs Glimepiride; The change from baseline to Week 52 is analyzed using analysis of ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of SBP (<130, ≥130 mmHg) at screening, and country as fixed effects and baseline body weight as a covariate; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LS Mean = -3.58, 95% CI 2-sided [-4.651 to -2.517], Standard Error of Mean 0.544

4. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) for Participants With SBP ≥130 mmHg at Week 12
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline, Week 12
Population: Analysis was performed on ITT population in participants with baseline SBP ≥130 mmHg. Missing data are imputed using washout imputation method.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Sotagliflozin 400 mg | Sotagliflozin 200 mg | Glimepiride
Number analyzed (Participants) | 79 | 161 | 81 | 175
mmHg | -5.34 (1.451) | -8.03 (1.064) | -9.12 (1.466) | -3.86 (1.081)
Statistical Analysis 1: Comparison: Sotagliflozin 400 mg vs Glimepiride; The change from baseline to Week 12 is analyzed using ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, and country as fixed effects, and baseline SBP as a covariate; Test type: Superiority; p = 0.0012, ANCOVA; Difference in LS Mean = -4.18, 95% CI 2-sided [-6.701 to -1.650], Standard Error of Mean 1.288
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0973, ANCOVA; Difference in LS Mean = -2.70, 95% CI 2-sided [-5.890 to 0.491], Standard Error of Mean 0.0973

5. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) for All Participants at Week 12
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline, Week 12
Population: ITT population included all randomized participants. Missing data are imputed using washout imputation method under the missing not at random framework.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Sotagliflozin 400 mg | Sotagliflozin 200 mg | Glimepiride
Number analyzed (Participants) | 159 | 317 | 160 | 318
mmHg | -2.64 (1.013) | -4.70 (0.791) | -4.77 (1.033) | -0.68 (0.795)
Statistical Analysis 1: Comparison: Sotagliflozin 400 mg vs Glimepiride; The change from baseline to Week 12 is analyzed using ANCOVA model with treatment groups, randomization strata of HbA1c (≤ 8.5, >8.5%) at screening, and country as fixed effects, and baseline SBP as a covariate; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LS Mean = -4.02, 95% CI 2-sided [-5.730 to -2.319], Standard Error of Mean 0.870

6. Secondary Outcome: Percentage of Participants With At Least One Documented Symptomatic Hypoglycemic Event
Description: Documented symptomatic hypoglycemia includes the typical symptoms of hypoglycemia (increased sweating, nervousness, asthenia/weakness, tremor, dizziness, increased appetite, palpitations, headache, sleep disorder, confusion, seizures, unconsciousness, and/or coma) and plasma glucose ≤ 70 mg/dL (3.9 mmol/L).
Time Frame: Up to Week 52
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sotagliflozin 400 mg | Sotagliflozin 200 mg | Glimepiride
Number analyzed (Participants) | 159 | 317 | 160 | 318
percentage of participants | 0.63 | 1.26 | 3.75 | 16.67
Statistical Analysis 1: Comparison: Sotagliflozin 400 mg vs Glimepiride; Weighted average of percentage difference between treatment groups from each stratum [randomization strata of HbA1c [≤8.5%, >8.5%] at screening, randomization strata of mean SBP [<130, ≥130 mmHg] at screening using Cochran-Mantel-Haenszel weights; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Percentage difference = -15.4, 95% CI 2-sided [-19.67 to -11.12]

7. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment.
Time Frame: Up to Week 52
Population: Safety population included all participants who had received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sotagliflozin 400 mg | Sotagliflozin 200 mg | Glimepiride
Number analyzed (Participants) | 159 | 317 | 159 | 317
percentage of participants | 57.2 | 59.9 | 56.6 | 49.2

8. Other Pre Specified Outcome: Percentage of Participants With Hypoglycemic Events
Description: Percentage of participants with hypoglycemic events are reported for the following 3 categories: Any hypoglycemia (as reported in the Electronic Case Report Form); Documented symptomatic hypoglycemia [typical symptoms of hypoglycemia (increased sweating, nervousness, asthenia/weakness, tremor, dizziness, increased appetite, palpitations, headache, sleep disorder, confusion, seizures, unconsciousness, and/or coma) and plasma glucose ≤ 70 mg/dL (3.9 mmol/L)]; Severe [an event requiring assistance of another person to actively administer carbohydrate, glucagon, intravenous glucose or other resuscitative actions] or documented symptomatic hypoglycemia [typical symptoms of hypoglycemia and plasma glucose ≤ 70 mg/dL].
Time Frame: Up to Week 52
Population: Safety population included all randomized participants who received at least 1 dose of double-blind investigational medicinal product (IMP) (regardless of the amount of treatment administered).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sotagliflozin 400 mg | Sotagliflozin 200 mg | Glimepiride
Number analyzed (Participants) | 159 | 317 | 159 | 317
percentage of participants
  Any hypoglycemia | 2.5 | 4.1 | 6.3 | 25.9
  Documented symptomatic hypoglycemia | 0.6 | 1.3 | 3.8 | 16.7
  Severe or documented symptomatic hypoglycemia | 0.6 | 1.3 | 3.8 | 16.7

ADVERSE EVENTS:
Time Frame: First dose of study drug to last dose of study drug (up to 52 weeks) + 2 weeks
Description: Safety population included all participants who had received at least one dose of study drug.
Arm/Group | Placebo | Sotagliflozin 400 mg | Sotagliflozin 200 mg | Glimepiride
All-Cause Mortality (participants affected / at risk) | 2/159 | 1/317 | 0/159 | 2/317
Serious Adverse Events (participants affected / at risk) | 11/159 | 17/317 | 11/159 | 14/317
Other Adverse Events (participants affected / at risk) | 30/159 | 49/317 | 21/159 | 22/317
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=159) | Sotagliflozin 400 mg (N=317) | Sotagliflozin 200 mg (N=159) | Glimepiride (N=317)
Acute left ventricular failure (Cardiac disorders) | 1 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Death (General disorders) | 1 | 0 | 0 | 0
Incarcerated hernia (General disorders) | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 1 | 0 | 0
Sudden cardiac death (General disorders) | 0 | 0 | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholecystitis infective (Infections and infestations) | 0 | 1 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 2
Pneumonia legionella (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis chronic (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Vascular graft stenosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebellar stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 0
Adnexa uteri mass (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=159) | Sotagliflozin 400 mg (N=317) | Sotagliflozin 200 mg (N=159) | Glimepiride (N=317)
Diarrhoea (Gastrointestinal disorders) | 11 | 14 | 8 | 7
Vulvovaginal mycotic infection (Infections and infestations) | 2 | 19 | 6 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 5 | 2 | 2
Headache (Nervous system disorders) | 11 | 14 | 7 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution must provide any proposed publication or presentation to Sponsor for Sponsor's review, comment and approval at least thirty (30) days prior to the proposed submission for publication date or the proposed presentation date. Sponsor shall have the right to have deleted from the final version of the publication any confidential information, proprietary information, or patentable subject matter.

DOCUMENTS (2):
  • Study Protocol (2018-04-11): https://cdn.clinicaltrials.gov/large-docs/71/NCT03332771/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/71/NCT03332771/SAP_001.pdf